CLINICAL TRIAL: NCT03488914
Title: Examining Community-based Effectiveness of a Substance Use and HIV Risk Reduction Intervention for Young Men of Color
Acronym: YMHP-CBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tyrel Starks, Associate Professor, Hunter College of City University of New York
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01DA041262 (NIH); R01DA041262 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Substance Use; Sexual Risk
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Randomization to YMHP or enhanced Treatment as Usual (eTAU)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): The YMHP intervention is a 4 session Motivational Interviewing (MI) intervention. In session 1, youth will choose which behavior to discuss first (substance use or sexual risk behavior), and the Health Educator counselor will elicit the client's view of the problem using standard MI techniques, building motivation for change by eliciting and reinforcing change talk, and clarifying the youth's own personal goals for maintaining their sexual health/considering changes in their substance use. The second session follows the same format for the second target behavior. In the subsequent two sessions, the counselor will discuss Pre-exposure Prophylaxis (PrEP) uptake as part of a change plan, continue to elicit and reinforce change talk, problem-solve barriers, consolidate commitment, and consider strategies to maintain behavior change.
  Interventions: Behavioral: YMHP Intervention
- Enhanced Treatment as Usual (Other): The Enhanced Treatment as Usual arm involves referring youth to standard of care services available at the community based organization for substance use and sexual health. This includes available services for Pre-exposure prophylaxis.
  Interventions: Behavioral: Enhanced Treatment as Usual

INTERVENTIONS:
Behavioral: YMHP Intervention
  Arms: Intervention
Behavioral: Enhanced Treatment as Usual
  Other Names: eTau
  Arms: Enhanced Treatment as Usual

SUMMARY:
This study will conduct an effectiveness trial of the 4-session evidence-based YMHP intervention for young men who have sex with men (YMSM) of color ages 15-29 at two CBOs in New York City, compared to usual care.

DETAILED DESCRIPTION:
We will conduct a comparative effectiveness trial (CET) with two intensities of treatment to be offered following field-based HIV counseling and testing (C&T) - the young men's health project (YMHP) intervention and an enhanced "treatment as usual" (eTAU) condition involving HIV prevention services provided at two community based organizations (CBOs) to test their relative effectiveness in reducing substance use and sexual risk behavior among HIV-negative YMSM. In collaboration with two CBOs, our goals are to better understand substance use and sexual health-related outcomes among HIV-negative YMSM who are unlikely to be treatment seeking and to implement the YMHP intervention in a way that will maximize portability and scalability. Working together with our collaborators will help to address practical problems at the frontline of service provision to pave the way for a comprehensive program to reduce substance use and HIV infection among YMSM.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative test result from the past 90 days
* 15-29 years of age
* Born biologically male or currently identifying as male
* Sex with men in the past 90 days
* ≥ 5 days of illicit drug use in the past 90 days
* ≥ 1 episode of condomless anal sex (CAS) in the past 90 days, or a positive sexually transmitted infection test result in the past 90 days.
* Living in the New York City area
* Able to communicate in English

Exclusion Criteria:

* Serious cognitive or psychiatric impairments
* ≥5 days of injection drug use in the past 90 days
* Currently taking Truvada as Pre-Exposure Prophylaxis (PrEP)

Ages: 15 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 86 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyrel J Starks, PhD, Principal Investigator — Hunter College, CUNY
Locations (2):
- United States (2):
  - Bridging Access to Care, Brooklyn, New York
  - BOOM!Health, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
Data sharing with scientific and health service community: We will have compiled structured de-identified datasets and can make them available for additional/secondary data analyses. It is our explicit intention that these data be readily accessible. We will collaborate with and make our data available to other researchers for additional/secondary analyses. Formal data sharing agreements will be developed to guide and encourage further data mining of the proposed datasets for various purposes.
Supporting Information: SAP
Time Frame: As per NIH policy
Access Criteria: The dissemination of any and all data collected under the NIH data sharing agreement will be released: a) In a timely manner following the time line of the project provide; and b) To the broader community, in accordance with NIH guidelines. Active dissemination to collaborators, community groups and through peer-reviewed articles will facilitate access to the data.

REFERENCES:
- [Derived] Coyle K, Carcone AI, Butame S, Pooler-Burgess M, Chang J, Naar S. Adapting the self-assessment of contextual fit scale for implementation of evidence-based practices in adolescent HIV settings. Implement Sci Commun. 2022 Oct 22;3(1):115. doi: 10.1186/s43058-022-00349-4. PMID 36273221
- [Derived] Bradford-Rogers J, Lopez-Matos J, Cain D, Lopez D, Starks TJ. Comparing the Efficiency of Online and Field-Based Outreach for the Recruitment of Black and Latino Sexual Minority Men into an HIV Prevention Implementation Trial. Prev Sci. 2022 Aug;23(6):900-906. doi: 10.1007/s11121-022-01367-3. Epub 2022 Apr 8. PMID 35394598
- [Derived] Parsons JT, Starks T, Gurung S, Cain D, Marmo J, Naar S. Clinic-Based Delivery of the Young Men's Health Project (YMHP) Targeting HIV Risk Reduction and Substance Use Among Young Men Who Have Sex with Men: Protocol for a Type 2, Hybrid Implementation-Effectiveness Trial. JMIR Res Protoc. 2019 May 21;8(5):e11184. doi: 10.2196/11184. PMID 31115346

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: The YMHP intervention is a 4 session Motivational Interviewing (MI) intervention. In session 1, youth will choose which behavior to discuss first (substance use or sexual risk behavior), and the Health Educator counselor will elicit the client's view of the problem using standard MI techniques, building motivation for change by eliciting and reinforcing change talk, and clarifying the youth's own personal goals for maintaining their sexual health/considering changes in their substance use. The second session follows the same format for the second target behavior. In the subsequent two sessions, the counselor will discuss Pre-exposure Prophylaxis (PrEP) uptake as part of a change plan, continue to elicit and reinforce change talk, problem-solve barriers, consolidate commitment, and consider strategies to maintain behavior change.
  YMHP Intervention
- Enhanced Treatment as Usual: The Enhanced Treatment as Usual arm involves referring youth to standard of care services available at the community based organization for substance use and sexual health. This includes available services for Pre-exposure prophylaxis.
  Enhanced Treatment as Usual
Period: Overall Study
Arm/Group | Intervention | Enhanced Treatment as Usual
Started | 47 | 39
Completed | 47 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Enhanced Treatment as Usual | Total
Number analyzed (Participants) | 47 | 39 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (3.37) | 24.3 (3.21) | 24.4 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 47 | 39 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 10 | 16 | 26
  Race/Ethnicity: Latino | 22 | 13 | 35
  Race/Ethnicity: White | 6 | 6 | 12
  Race/Ethnicity: Other | 9 | 4 | 13
Site [Count of Participants; unit: Participants] — Participants were enrolled at two different study sites. Site names have been de-identified.
  Participants
    Study Site 1 | 33 | 11 | 44
    Study Site 2 | 14 | 28 | 42
Relationship Status [Count of Participants; unit: Participants]
  Single | 37 | 25 | 62
  Partnered | 10 | 14 | 24
Education [Count of Participants; unit: Participants]
  4-Year College Degree | 7 | 6 | 13
  Less than 4-Year Degree | 26 | 21 | 47
  Missing | 14 | 12 | 26
Employment [Count of Participants; unit: Participants]
  Part-time | 9 | 12 | 21
  Full-time | 7 | 6 | 13
  Missing | 31 | 21 | 52

OUTCOME MEASURES:

1. Primary Outcome: Illicit Drug Use Days
Description: The self-reported number of illicit drug use days (not including marijuana) in the past 90 days
Time Frame: Baseline, 3-Month, 6-Month, 9-Month, 12-Month, 15-Month
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Enhanced Treatment as Usual
Number analyzed (Participants) | 47 | 39
days
  Baseline | 3.04 (7.05) | 11.62 (6.04)
  3-Month | 2.00 (5.03) | 6.04 (11.10)
  6-Month | 1.19 (2.97) | 6.29 (12.48)
  9-Month | 3.81 (8.19) | 3.77 (9.08)
  12-Month | 2.00 (4.83) | 4.35 (11.37)
  15-Month | 2.08 (5.25) | 6.19 (11.30)
Statistical Analysis 1: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .19, negative binomial regression; Model testing whether condition predicted illicit drug use days at 3-months; Slope = -1.09, 95% CI 2-sided [-2.78 to .56]
Statistical Analysis 2: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .12, negative binomial regression; Model testing whether condition predicted illicit drug use days at 6-months; negative binomial regression = -1.66, 95% CI 2-sided [-3.78 to .48]
Statistical Analysis 3: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .99, negative binomial regression; Model testing whether condition predicted illicit drug use days at 9-months; Slope = .01, 95% CI 2-sided [-2.05 to 2.07]
Statistical Analysis 4: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .42, negative binomial regression; Model testing whether condition predicted illicit drug use days at 12-months; Slope = -.78, 95% CI 2-sided [-2.67 to 1.11]
Statistical Analysis 5: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .18, negative binomial regression; Model testing whether condition predicted illicit drug use days at 15-months; Slope = -1.09, 95% CI 2-sided [-2.69 to .51]

2. Primary Outcome: Condomless Anal Sex Acts
Description: The self-reported number of condomless anal sex acts with male partners in the past 90 days
Time Frame: Baseline, 3-Month, 6-Month, 9-Month, 12-Month, 15-Month
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: acts
Arm/Group | Intervention | Enhanced Treatment as Usual
Number analyzed (Participants) | 47 | 39
acts
  Baseline | 10.38 (13.02) | 14.36 (15.59)
  3-Months | 9.71 (17.5) | 9.47 (14.88)
  6-Months | 3.38 (5.16) | 11.14 (16.49)
  9-Months | 12.45 (15.28) | 10.92 (16.01)
  12-Months | 7.3 (10.32) | 6.88 (11.83)
  15-Months | 6.56 (9.02) | 10 (11.99)
Statistical Analysis 1: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .96, negative binomial regression; Model testing whether condition predicted condomless anal sex acts at 3-months; Slope = .03, 95% CI 2-sided [-.86 to .99]
Statistical Analysis 2: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .03, negative binomial regression; Model testing whether condition predicted condomless anal sex acts at 6-months; Slope = -1.19, 95% CI 2-sided [-2.25 to -.14]
Statistical Analysis 3: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .79, negative binomial regression; Model testing whether condition predicted condomless anal sex acts at 9-months; Slope = .13, 95% CI 2-sided [-.83 to 1.10]
Statistical Analysis 4: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .91, negative binomial regression; Model testing whether condition predicted condomless anal sex acts at 12-months; Slope = .06, 95% CI 2-sided [-.99 to 1.11]
Statistical Analysis 5: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .44, negative binomial regression; Model testing whether condition predicted condomless anal sex acts at 15-months; Slope = -.42, 95% CI 2-sided [-1.50 to .65]

3. Primary Outcome: Marijuana Use Days
Description: The self-reported number of marijuana use days in the past 90 days
Time Frame: Baseline, 3-Month, 6-Month, 9-Month, 12-Month, 15-Month
Population: intent-to-treat population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Enhanced Treatment as Usual
Number analyzed (Participants) | 47 | 39
days
  Baseline | 33.11 (32.59) | 46.15 (36.14)
  3-Months | 34.19 (36.97) | 44.39 (42.45)
  6-Months | 35.81 (39.4) | 24.50 (32.86)
  9-Months | 32.52 (35.26) | 42 (39.57)
  12-Months | 37.75 (36.93) | 29.24 (39.22)
  15-Months | 25.08 (32.64) | 36.06 (40.25)
Statistical Analysis 1: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .54, negative binomial regression; Model testing whether condition predicted marijuana use days at 3-months; Slope = -.26, 95% CI 2-sided [-1.09 to .58]
Statistical Analysis 2: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .49, negative binomial regression; Model testing whether condition predicted marijuana use days at 6-months; Slope = .38, 95% CI 2-sided [-.70 to 1.46]
Statistical Analysis 3: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .59, negative binomial regression; Model testing whether condition predicted marijuana use days at 9-months; Slope = -.26, 95% CI 2-sided [-1.18 to .66]
Statistical Analysis 4: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .65, negative binomial regression; Model testing whether condition predicted marijuana use days at 12-months; Slope = .26, 95% CI 2-sided [-.86 to 1.37]
Statistical Analysis 5: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .49, negative binomial regression; Model testing whether condition predicted marijuana use days at 15-months; Slope = -.36, 95% CI 2-sided [-1.40 to .67]

4. Secondary Outcome: Alcohol Use Days
Description: The self-reported number of alcohol use days in the past 90 days
Time Frame: Baseline, 3-Month, 6-Month, 9-Month, 12-Month, 15-Month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Enhanced Treatment as Usual
Number analyzed (Participants) | 47 | 39
days
  Baseline | 20.26 (22.15) | 30.10 (27.14)
  3-Months | 18.81 (26.42) | 27.04 (28.57)
  6-Months | 9.94 (11.64) | 20.29 (21.88)
  9-Months | 16.08 (20.98) | 27.31 (21.76)
  12-Months | 14.45 (18.72) | 18.53 (21.16)
  15-Months | 11.35 (14.05) | 17.75 (20.52)
Statistical Analysis 1: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .31, negative binomial regression; Model testing whether condition predicted alcohol use days at 3-months; Slope = -.36, 995% CI 2-sided [-1.07 to .34]
Statistical Analysis 2: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .10, negative binomial regression; Model testing whether condition predicted alcohol use days at 6-months; Slope = -.71, 95% CI 2-sided [-1.57 to .15]
Statistical Analysis 3: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .20, negative binomial regression; Model testing whether condition predicted alcohol use days at 9-months; Slope = -.53, 95% CI 2-sided [-1.34 to .28]
Statistical Analysis 4: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .58, negative binomial regression; Model testing whether condition predicted alcohol use days at 12-months; Slope = -.25, 95% CI 2-sided [-1.14 to .64]
Statistical Analysis 5: Comparison: Intervention vs Enhanced Treatment as Usual; Test type: Superiority; p = .34, negative binomial regression; Model testing whether condition predicted alcohol use days at 15-months; Slope = -.45, 95% CI 2-sided [-1.37 to .47]

ADVERSE EVENTS:
Time Frame: 15-months
Arm/Group | Intervention | Enhanced Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/39
Other Adverse Events (participants affected / at risk) | 0/47 | 0/39

LIMITATIONS AND CAVEATS:
Enrollment was delayed substantially by implementation challenges early in the trial. Due to the COVID pandemic, enrollment closed early. As a result, the sample enrolled was less than half of the original proposal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03488914/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT03488914/ICF_001.pdf